CLINICAL TRIAL: NCT00388843
Title: Short Term Carotid Plaque Regression in Patients With Atherosclerotic Disease Taking Statins Assessed by High Field MRI
Brief Title: Carotid Plaque Regression With Statin Treatment Assessed by High Field Magnetic Resonance Imaging (MRI)
Status: Withdrawn | Type: Observational
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Raymond Q. Migrino, Department of Medicine, Medical College of Wisconsin
Other Study IDs: PRO00002285
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Carotid Atherosclerosis
Keywords: carotid atherosclerosis; magnetic resonance imaging; atherosclerosis; ultrasound; inflammation; statins; vulnerable plaque; stroke
MeSH Terms: conditions — Carotid Artery Diseases; Atherosclerosis; Inflammation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dose Increased: Patients presenting with symptoms of coronary artery disease or stroke/suspected stroke, with carotid plaque > 1.1 mm, and whose statin dose is increased to moderate to high dose by their clinicians.
- Dose Maintained: Patients presenting with symptoms due to coronary artery disease or stroke/suspected stroke, with carotid plaque > 1.1 mm, on no statins or whose statin dose was unchanged by their clinicians.

SUMMARY:
The purpose of the study is to determine if short term (6 months) treatment with statins to lower low-density lipoprotein (LDL) in vascular disease patients with carotid plaque will be associated with a measurable reduction in carotid plaque volume using 3 Tesla MRI. The researchers will correlate the change in plaque volume to degree of LDL lowering. The researchers will also study if brief treatment will lead to change in plaque composition. The researchers will compare the change in plaque volume measured by 3T MRI with plaque burden measured by ultrasound.

DETAILED DESCRIPTION:
Atherosclerotic vascular disease is the leading cause of death in the United States. Atherosclerosis develops with increasing plaque burden and eccentric arterial wall expansion or remodeling, later leading to luminal obstruction. More than 90% of patients with CAD have carotid plaques. Statins have been shown to cause plaque regression in the carotid and coronary arteries. However, there is ongoing controversy about how low the target LDL should be in atherosclerotic patients. The benefits of aggressive LDL lowering with higher statin doses are counterbalanced by the potential for liver and muscle toxicity. High field (3 Tesla) MRI is a promising new modality for measuring plaque volume with high spatial resolution. It is not clear whether increasing statin dose will lead to plaque volume reduction in the short-term (6 months) that can be measured by this new modality.

The primary aim of the study is to determine if LDL lowering using statins in vascular disease patients with carotid plaque will be associated with measurable reduction in carotid plaque volume in the short term (6 months) using 3T MRI.

The four secondary aims of the study are as follows:

To compare the short term carotid plaque volume change using high field MRI in vascular disease patients whose statin dose was increased (dose increased) versus those whose statin dose was maintained (dose maintained).

To determine if increasing statin dose in patients with carotid plaque will lead to measurable change in carotid plaque composition in the short term (6 months) using 3T MRI.

To compare the carotid plaque volume change using 3T MRI with change in plaque burden score using carotid ultrasound .

To determine the relationship between change in plaque volume with change in lipid levels (total cholesterol, LDL, HDL) and change in inflammatory markers (cytokines, high sensitivity CRP).

The study is significant because it will provide insight into optimal statin treatment for atherosclerotic disease. It will also test a new modality for measurement of plaque burden. A reliable and sensitive test with high spatial resolution that accurately measures change in plaque volume will be helpful in assessing response to treatment and as a tool for future clinical trials in assessing efficacy of new treatment modalities that may reduce the need for expensive, long term studies that rely on clinical events for outcome measurement.

ELIGIBILITY:
Inclusion criteria:

* Adult (> 21 years old) patients.
* Diagnosed with coronary artery disease or suspected cerebrovascular accident.
* For dose increased subjects, patients whose statin dose or LDL lowering therapy is doubled or increased from standard dose to high dose (see table).
* For dose maintained subjects, patients whose statin dose or LDL lowering therapy is maintained at standard dose (see table).
* Standard Dose (reported LDL↓ < 40% from literature)

  * Drug Daily Dose/s: (md/day)
  * atorvastatin 10
  * simvastatin 5, 10, 20
  * pravastatin 10, 20, 40, 80
  * fluvastatin 20, 40, 80
  * lovastatin 10, 20, 40
* High Dose (reported LDL↓ > 40% from literature)

  * Drug Daily Dose/s (mg/day)
  * atorvastatin 40, 80
  * simvastatin 40, 80
  * lovastatin 80
  * rosuvastatin 5, 10, 20, 40
  * Addition of non-statin lipid transfer (tx) (e.g., ezetimibe, fibrate, niacin) to standard statin dose

Exclusion criteria:

* severe claustrophobia causing inability to undergo MRI implanted ferromagnetic materials (pacemakers, defibrillators, TENS units, aneurysm clips, etc.) that are not suitable for MRI in the clinical setting
* patients anticipated to undergo carotid stenting or surgery in next 6 months
* patients unable to lie flat for 1 hour
* patients requiring supplemental oxygen
* pregnant women
* patients who could not be followed up for 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with coronary artery disease or suspected cerebrovascular accident who have carotid plaque (> 1.1 mm) and whose statin dose has been increased to moderate or high dose (increased statin dose) or maintained (maintained statin dose).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in carotid artery plaque volume assessed by carotid MRI at 6 months | 6 months

SECONDARY OUTCOMES:
Change in carotid intima media thickness on ultrasound at 6 months | 6 months
Change in plaque composition by carotid MRI at 6 months | 6 months
Change in inflammatory markers at 6 months | 6 months
Change in regional wall shear stress in the carotid artery | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Migrino, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Memorial and Lutheran Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- See also: Medical College of Wisconsin site — http://www.mcw.edu